CLINICAL TRIAL: NCT00005347
Title: Framingham Cycle V Offspring-Spouse Nutrition Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4216; R01HL046193 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension; Obesity; Diabetes Mellitus; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension; Obesity; Diabetes Mellitus; Atherosclerosis

SUMMARY:
To examine the associations between diet, nutrition and coronary heart disease (CHD) incidence over seven years using the Cycle V Framingham Offspring/Spouse examination ; to examine the cross-sectional associations between dietary variables and major cardiovascular disease risk factors, to examine changes in dietary behaviors and their determinants over seven years; and to characterize the influences of dietary behavior changes on risk factor status between 1984-88 and 1991-94.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The data collection efforts and cross-sectional analyses were carried out among approximately 3800 males and females during the scheduled 1991-1994 Cycle V Framingham Offspring/Spouse study. The secular trend and longitudinal analyses also included data that were collected during the Cycle III Offspring/Spouse studies in 1984-88. Of particular interest were dietary variables which play a major role in serum total cholesterol and lipoprotein regulation. Additional dietary variables which were associated with major cardiovascular risk factors ((elevated) blood pressure, glucose (in)tolerance, (excess) body weight or physical (in)activity, and smoking) or that may predict CHD endpoints were included in the analyses. The potential confounding effects or interactions between dietary and risk factor variables were considered. Separate analyses were carried out in males and females.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-02; Study Completion 1997-01 (Actual)

REFERENCES:
- [Background] Drach GW. Urinary lithiasis. J Urol. 1980 Mar;123(3):348. doi: 10.1016/s0022-5347(17)55928-5. No abstract available. PMID 7359634
- [Background] Posner BM, Franz MM, Quatromoni PA, Gagnon DR, Sytkowski PA, D'Agostino RB, Cupples LA. Secular trends in diet and risk factors for cardiovascular disease: the Framingham Study. J Am Diet Assoc. 1995 Feb;95(2):171-9. doi: 10.1016/S0002-8223(95)00043-7. PMID 7852683